CLINICAL TRIAL: NCT06981832
Title: Physical Activity for Haemodialysis Patients: Evaluation of Personalised Support by an Adapted Physical Activity Teacher and an Advanced Practice Nurse
Acronym: HE-MOVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Departemental Vendee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CHD25_0004
Record Dates: First submitted 2025-05-13; First posted 2025-05-21 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Hemodialysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personalised support (advanced practice nurse and adapted physical activity teacher) (Experimental)
  Interventions: Behavioral: Personalised support (advanced practice nurse and adapted physical activity teacher)
- Standard support (advanced practice nurse) (Active Comparator)
  Interventions: Behavioral: Standard support (advanced practice nurse)

INTERVENTIONS:
Behavioral: Personalised support (advanced practice nurse and adapted physical activity teacher) — Personalised support (advanced practice nurse and adapted physical activity teacher)
  Arms: Personalised support (advanced practice nurse and adapted physical activity teacher)
Behavioral: Standard support (advanced practice nurse) — Standard support (advanced practice nurse)
  Arms: Standard support (advanced practice nurse)

SUMMARY:
Physical activity is defined as 'any bodily movement produced by skeletal muscles that results in an energy expenditure greater than that of the resting metabolism'. Physical activity includes 'activities of daily living, physical exercise and sporting activities'.

The scientific community is agreed in recognising the benefits of physical activity, both in healthy individuals and in those suffering from chronic diseases.

With this in mind, the law of 2 March 2022 allows doctors to prescribe Adapted Physical Activity.

In the case of chronic renal failure, there are a number of factors that can limit physical activity in haemodialysis patients, such as anaemia, nutritional status and post-dialysis fatigue.

However, the risks associated with a sedentary lifestyle play a role in the development of chronic disease, in particular hypertension and diabetes. The benefits of physical activity have been widely identified in chronic renal failure, particularly in terms of cardiovascular and muscular function.

More generally, physical activity has a positive impact on physical, psychological and social quality of life (increase in overall quality of life score, improved sleep, reduced pain, etc.).

Physical activity should therefore be encouraged in patients with chronic renal failure, whether on dialysis or not, whatever their age.

The aim of this study is to assess whether individualised support (from an advanced practice nurse and an adapted physical activity teacher) improves the practice of physical activity at home in patients who have been on haemodialysis for less than a year, and whether this improvement is sustainable over time.

ELIGIBILITY:
Pre-Inclusion Criteria:

* Patient over 18 years of age
* Patient who has been receiving haemodialysis for less than a year
* Patient with medical prescription for physical activity
* Patient able to understand the protocol and having given consent to participate in the research,
* Patient affiliated to the social security system or entitled beneficiary

Inclusion Criteria:

* Patient with physical activity considered low or moderate according to the IPAQ questionnaire

Exclusion Criteria:

* Patients with medical contraindications to adapted physical activity
* Patients with a lower limb amputation
* Patients undergoing peritoneal dialysis
* Patient with a peritoneal dialysis project
* Patient participating in another clinical research protocol with an impact on the research objectives
* Patient already randomised in the study
* Patient who is pregnant, parturient, breastfeeding or able to procreate without effective contraception at the time of inclusion*.
* Patients under guardianship, curatorship or deprived of liberty
* Patient under activated future protection mandate
* Patient under family habilitation
* Patient under court protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-10-28 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Patients with a level of physical activity considered moderate or high, assessed using the physical activity questionnaire (IPAQ) 6 months after the start of the intervention | 6 months after the start of the intervention
  The level of physical activity according to the IPAQ questionnaire is defined as follows:
  1. - Low
     * No activity is reported OR
     * Some activity is reported but without reaching levels 2 or 3.
  2. - Moderate Corresponds to one of the following 3 criteria:
     * 3 or more days of intense activity lasting at least 20 minutes a day OR
     * 5 days or more of moderate intensity activity and/or walking for at least 30 minutes a day OR
     * 5 days or more of activity combining walking, moderate or high intensity activities, thus achieving at least 600 MET-minutes/week.
  3. - High Corresponds to one of the 2 following criteria:
     * Intense activity on at least 3 days a week, achieving at least 1500 MET-minutes/week OR
     * 7 or more days of activity combining walking and moderate or high-intensity activities, achieving at least 3000 MET-minutes/week.

CONTACTS AND LOCATIONS:
Overall Officials: Emilie VINCENT, Principal Investigator — Centre H
Locations (1):
- Centre Hospitalier Departemental Vendée, La Roche-sur-Yon, France

IPD SHARING:
Plan to Share IPD: No